CLINICAL TRIAL: NCT04871685
Title: ECOVITA Study. Observational Study on Sars-COV 2 Population Hospitalized in the Italian Country
Brief Title: The ECOVITA Study - Validation of LUS Score in SARS-CoV-2 Disease, i.e COVID-19
Acronym: ECOVITA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Luca Rinaldi, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: Vanvitelli
Record Dates: First submitted 2021-04-27; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: lung ultrasound
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Covid Center UOC Vanvitelli, Naples: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Cotugno Hospital, Naples: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center "Del Mare Hospital", Naples: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Santa Maria delle Grazie Hospital, Pozzuoli: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Monaldi Hospital, Naples: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Vannini Hospital, Rome: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Bassini Hospital, ASST Milano Nord: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Melfi Hospital: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound
- Covid Center Messina University Hospital: Patients hospitalized due to Sars-Cov-2 disease either in emergency or ordinary medicine/intensive care units
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — the patients underwent to a non invasive diagnostic exam to identify and monitor clinical conditions and onset of respiratory complications due to COVID-19

SUMMARY:
Lung Ultrasound (LUS) has been revealing an extremely useful tool to identify and monitor complications from Sars-COV-2 disease. Recently, a research group has proposed a score, named LUS Score, able to optimize the use of this diagnostic technique. LUS Score is computed analyzing chest posterior and lateral spaces, considering the number of artefacts generated by the inflammed interstitium (B lines), the characteristics of the pleural line and the presence or not of consolidation areas.

The comparison between LUS and chest tomography (CT), the current gold standard for the diagnosis of interstitial pneumonia by COVID-19, has confirmed from the preliminary data, the reliability of such technique. Hence, the validation on a really large sample size of the ultrasound tool performed by dedicated personnel with high expertise, may allow the validation both in the clinical practice and in emergency and ordinary wards.

ELIGIBILITY:
Inclusion Criteria:

* men and women;
* confirmed COVID19 diagnosis after nasal-oropharyngeal swab;
* any symptom at hospitalization
* any therapy
* any pre-existing comorbidity

Exclusion Criteria:

* pregnant women
* healthy subjects with other respiratory diseases different from COVID-19

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized due to COVID19 infection
Sampling Method: Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-05-03 (Estimated)

PRIMARY OUTCOMES:
validation of lung ultrasound score | 6 months
  validation of lung ultrasound in the clinical practice of diagnosis of complications of low respiratory tracts during COVID-19

SECONDARY OUTCOMES:
Association of LUS score with clinical outcome | 6 months
  assessment of LUS score association with the clinical course of disease (final outcome, either discharged or in-hospital mortality
Association of LUS score with duration of hospitalization (days) | 6 months
  assessment of LUS score association with hospitalization days
Association of LUS score with respiratory support required | 6 months
  assessment of LUS score association with requirement of either sub-intensive or intensive therapy)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No